CLINICAL TRIAL: NCT04256343
Title: The Sensitivity of Differing D2O Dosing Strategies and Mass Spectrometry-based Analytical Techniques to Determine Rates of Muscle Protein Synthesis in Young Men and Women
Brief Title: D2O Dosing Strategies to Assess Muscle Protein Synthesis
Acronym: D2O-MPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID and lack of funding
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 8300
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2020-02

CONDITIONS: Hypertrophy
Keywords: Muscle; Muscle protein synthesis; Deuterium
MeSH Terms: conditions — Hypertrophy | interventions — Deuterium Oxide

STUDY DESIGN:
Intervention Model Description: This study will be a double blind, randomized, parallel control trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the outcomes assessors will be blinded to which dose of D2O the participant received, only the lead principal investigator and the investigators will know which condition each participant has been assigned to. The protein synthesis analysis will be carried out in a blinded fashion such that the individuals utilizing the analytical machines/interpreting the data will be unaware of who was assigned to which condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D2O Dose 1 (Experimental): Lower dose of D2O for MPS
  Interventions: Other: Deuterium Oxide (D2O) Dose
- D2O Dose 2 (Experimental): Moderate dose of D2O MPS
  Interventions: Other: Deuterium Oxide (D2O) Dose
- D2O Dose 3 (Experimental): Higher dose of D2O for MPS
  Interventions: Other: Deuterium Oxide (D2O) Dose

INTERVENTIONS:
Other: Deuterium Oxide (D2O) Dose — 1 of 3 differing deuterium oxide (D2O) doses will provided to each of the participants to be consumed daily to assess muscle protein synthesis.

SUMMARY:
Skeletal muscle mass is regulated by the balance of muscle protein synthesis (MPS) and muscle protein breakdown (MPB). MPS is sensitive to exogenous stimuli, particularly exercise and protein ingestion. Much of what the investigators currently know about the impact of exercise and protein feeding on MPS has been derived from acute stable isotopic tracers in a controlled laboratory setting. However, recently, the field of skeletal muscle protein metabolism has moved towards the use of deuterium oxide (deuterated water (D2O)) to measure MPS. The ease of administration and the scope to measure turnover in a range of substrates whilst negating the need for strictly controlled laboratory settings makes D2O the ideal candidate to provide a more holistic view of in vivo skeletal muscle metabolism.

DETAILED DESCRIPTION:
Currently, there is a lack of consensus amongst researchers regarding the dosing strategies of D2O provision for measuring fraction-specific (myofibrillar, mitochondrial and sarcoplasmic) protein synthetic rates. In addition, the analytical equipment (i.e., mass spectrometers) required to carry out the analysis of skeletal muscle-bound alanine are technically challenging, offer varying degrees of sensitivity that may drastically influence outcome measures and the expense of analysis differs greatly between the type of mass spectrometer required.Thus, this study will employ different D2O doses to assess basal and exercise plus protein feeding-induced rates of acute and integrated MPS in healthy young men and women. This will provide researchers with insight into the amount of D2O required to accurately assess MPS and the sensitivity of the analytical machine employed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, between the ages of 18 - 35 years (inclusive)
2. Have a body mass index (BMI) between 18-30 kg·m2 (inclusive)
3. Be in general good health as assessed by a general health questionnaire
4. Non-smoking
5. Willing and able to provide informed consent

Exclusion Criteria:

1. Ingestion of deuterated water (D2O) in the previous ~6 months.
2. Routine/daily usage of non-steroidal anti-inflammatory drugs (NSAIDS, prescription use or daily use of over the counter medication), use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), any anabolic steroid, creatine, whey protein supplements, casein or branched-chain amino acids (BCAAs) within 45 days prior to screening.
3. Use of tobacco or related products.
4. Veganism or vegetarianism
5. Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements.
6. Use assistive walking devices (e.g., cane or walker)
7. History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
8. Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude oral protein supplement ingestion and/or assessment of safety and study objectives.
9. Any cachexia-related condition (e.g., relating to cancer, tuberculosis or human immunodeficiency virus infection and acquired immune deficiency syndrome) or any genetic muscle diseases or disorders
10. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing)
11. Hypersensitivity or known allergy to any of the components in the test formulations.
12. Excessive alcohol consumption (>21 units/week)
13. History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy (up to 81mg of baby aspirin per day taken as a prophylactic is permitted).
14. History of statin myalgia.
15. Personal or family history of clotting disorder or deep vein thrombosis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis | 7 days
  this study will employ different D2O doses to assess basal and exercise plus protein feeding-induced rates of acute and integrated MPS in healthy young men and women.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, Ph.D., Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No